CLINICAL TRIAL: NCT05129475
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, 2 SEQUENCE, 2 PERIOD CROSSOVER STUDY TO EVALUATE THE EFFECT OF HIGH-FAT MEAL ON THE RELATIVE BIOAVAILABILITY OF PF-07321332 BOOSTED WITH RITONAVIR IN HEALTHY ADULT PARTICIPANTS
Brief Title: Food Effect Study to Evaluate the Effect of High-Fat Meal on the Relative Bioavailability of PF-07321332 Boosted With Ritonavir in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671019
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2022-12

CONDITIONS: Healthy Participants
Keywords: food effect; COVID-19 (Coronavirus disease 2019); SARS-CoV (severe acute respiratory syndrome coronavirus)
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — nirmatrelvir and ritonavir drug combination; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Single oral dose of ritonavir at -12 hours prior to PF-07321332/ritonavir dosing, followed by single oral dose of PF-07321332/ritonavir under fasted conditions. Ritonavir will continue to be dosed at 12 hours PF-07321332 dosing.
  Interventions: Drug: PF-07321332/ritonavir; Drug: Ritonavir
- Treatment B (Experimental): Single oral dose of ritonavir at -12 hours prior to PF 07321332/ritonavir dosing, followed by single oral dose of PF-07321332/ritonavir under fed conditions. Ritonavir will continue to be dosed at 12 hours PF-07321332 dosing.
  Interventions: Drug: PF-07321332/ritonavir; Drug: Ritonavir

INTERVENTIONS:
Drug: PF-07321332/ritonavir — Single oral dose of PF-07321332 300 mg (2 × 150 mg tablets)/ritonavir 100 mg under fed or fasted conditions at 0 hour on Day 1
Drug: Ritonavir — Single oral dose of ritonavir 100 mg at -12 hours prior to PF-07321332/ritonavir dosing, and ritonavir 100 mg will be dosed at 12 hours after PF-07321332/ritonavir dosing.

SUMMARY:
This is a Phase 1, open label, single dose, randomized, 2-treatment, 2-sequence, 2-period crossover study to evaluate the effect of high-fat meal on the relative bioavailability of PF-07321332 boosted with ritonavir following single dose oral administration of PF-07321332 in combination with ritonavir using 150 mg tablet formulation of PF-07321332 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECGs. Female participants of childbearing potential must have a negative pregnancy test.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Positive test result (RT-PCR) for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy- or brady brady-arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg,. contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sagawa K, Lin J, Jaini R, Di L. Physiologically-Based Pharmacokinetic Modeling of PAXLOVID with First-Order Absorption Kinetics. Pharm Res. 2023 Aug;40(8):1927-1938. doi: 10.1007/s11095-023-03538-5. Epub 2023 May 25. PMID 37231296
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 healthy participants signed the informed consent form (ICF) and were enrolled in the study. All of them received the study treatment.
Groups:
- PF-07321332 Fasted + Ritonavir Then PF-07321332 Fed + Ritonavir: Period 1: Participants received a single oral dose of PF-07321332 300 milligram (mg) (2 tablets of 150 mg each) on Day 1 and 3 doses of ritonavir 100 mg at -12 hour (Day -1), 0 hour and 12 hour (Day 1) related to PF-07321332 dosing under fasted conditions in Period 1 and serial pharmacokinetic (PK) samples were collected up to 48 hours post dose (study Day 3). Period 2: Period 2 started on study Day 4 (Day -1 of Period 2). Participants received a single oral dose of PF-07321332 300 mg on Day 1 (study Day 5) and 3 doses of ritonavir 100 mg at -12 hour (Day -1), 0 hour and 12 hour (Day 1) related to PF-07321332 dosing under fed conditions and PK samples collected up to 48 hours post dose (study Day 7). A minimum of 4 days washout period was present between the PF-07321332 dosing of Period 1 and Period 2. Participants were followed up to maximum of 35 days after the last administration of study drug.
- PF-07321332 Fed + Ritonavir Then PF-07321332 Fasted + Ritonavir: Period 1: Participants received a single oral dose of PF-07321332 300 mg (2 tablets of 150 mg each) on Day 1 and 3 doses of ritonavir 100 mg at -12 hour (Day -1), 0 hour and 12 hour (Day 1) related to PF-07321332 dosing under fed conditions in Period 1 and serial PK samples were collected up to 48 hours post dose (study Day 3). Period 2: Period 2 started on study Day 4 (Day -1 of Period 2). Participants received a single oral dose of PF-07321332 300 mg on Day 1 (study Day 5) and 3 doses of ritonavir 100 mg at -12 hour (Day -1) , 0 hour and 12 hour (Day 1) related to PF-07321332 dosing under fasted conditions and PK samples collected up to 48 hours post dose (study Day 7). A minimum of 4 days washout period was present between the PF-07321332 dosing of Period 1 and Period 2. Participants were followed up to maximum of 35 days after the last administration of study drug.
Period: Period 1
Arm/Group | PF-07321332 Fasted + Ritonavir Then PF-07321332 Fed + Ritonavir | PF-07321332 Fed + Ritonavir Then PF-07321332 Fasted + Ritonavir
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | PF-07321332 Fasted + Ritonavir Then PF-07321332 Fed + Ritonavir | PF-07321332 Fed + Ritonavir Then PF-07321332 Fasted + Ritonavir
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | PF-07321332 Fasted + Ritonavir Then PF-07321332 Fed + Ritonavir | PF-07321332 Fed + Ritonavir Then PF-07321332 Fasted + Ritonavir
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- PF-07321332 Fasted + Ritonavir Then PF-07321332 Fed + Ritonavir: Period 1: Participants received a single oral dose of PF-07321332 300 mg (2 tablets of 150 mg each) on Day 1 and 3 doses of ritonavir 100 mg at -12 hour (Day -1), 0 hour and 12 hour (Day 1) related to PF-07321332 dosing under fasted conditions in Period 1 and serial PK samples were collected up to 48 hours post dose (study Day 3). Period 2: Period 2 started on study Day 4 (Day -1 of Period 2). Participants received a single oral dose of PF-07321332 300 mg on Day 1 (study Day 5) and 3 doses of ritonavir 100 mg at -12 hour (Day -1), 0 hour and 12 hour (Day 1) related to PF-07321332 dosing under fed conditions and PK samples collected up to 48 hours post dose (study Day 7). A minimum of 4 days washout period was present between the PF-07321332 dosing of Period 1 and Period 2. Participants were followed up to maximum of 35 days after the last administration of study drug.
- Total: Total of all reporting groups
Arm/Group | PF-07321332 Fasted + Ritonavir Then PF-07321332 Fed + Ritonavir | PF-07321332 Fed + Ritonavir Then PF-07321332 Fasted + Ritonavir | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (13.06) | 40.2 (13.03) | 46.9 (14.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 3 | 2 | 5
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-07321332
Description: Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration was determined by linear/log trapezoidal method and reported in this outcome measure.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: The PK parameter analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Groups:
- PF-07321332 300 mg/Ritonavir 100 mg Fed: Participants received a single oral dose of PF-07321332 300 mg on Day 1 and 3 doses of 100 mg ritonavir at -12 hours (Day -1), 0 hours and 12 hours (Day 1) related to PF-07321332 dosing in either Period 1 or Period 2 under fed conditions. Participants were followed up to maximum of 35 days after the last dose of study drug.
- PF-07321332 300 mg/Ritonavir 100 mg Fasted: Participants received a single oral dose of PF-07321332 300 mg on Day 1 and 3 doses of 100 mg ritonavir at -12 hours (Day -1), 0 hours and 12 hours (Day 1) related to PF-07321332 dosing in either Period 1 or Period 2 under fasted conditions. Participants were followed up to maximum of 35 days after the last dose of study drug.
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Nanogram*hour per milliliter | 43360 (31) | 35860 (35)
Statistical Analysis 1: Comparison: PF-07321332 300 mg/Ritonavir 100 mg Fed vs PF-07321332 300 mg/Ritonavir 100 mg Fasted; Test type: Other; Ratio of Adjusted Geometric Means = 120.90, 90% CI 2-sided [109.30 to 133.74] — Analysis done using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Ratio and 90% CI are expressed as percentages

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07321332
Description: AUCinf was calculated by AUClast + (Clast/kel). AUClast was the area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast). Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Nanogram*hour per milliliter | 44050 (31) | 36810 (36)
Statistical Analysis 1: Comparison: PF-07321332 300 mg/Ritonavir 100 mg Fed vs PF-07321332 300 mg/Ritonavir 100 mg Fasted; Test type: Other; Ratio of Adjusted Geometric Means = 119.67, 90% CI 2-sided [108.75 to 131.68] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07321332
Description: Cmax was defined as maximum observed plasma concentration. It was observed directly from data.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Nanogram per milliliter | 5951 (31) | 3696 (44)
Statistical Analysis 1: Comparison: PF-07321332 300 mg/Ritonavir 100 mg Fed vs PF-07321332 300 mg/Ritonavir 100 mg Fasted; Test type: Other; Ratio of Adjusted Geometric Means = 161.01, 90% CI 2-sided [139.05 to 186.44] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07321332
Description: Tmax was defined as the time to reach maximum observed plasma concentration of PF-07321332.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Hours | 2.50 [1.50 to 4.00] | 2.29 [1.00 to 3.00]

5. Secondary Outcome: Terminal Elimination Half-life (t1/2) of PF-07321332
Description: t1/2 was calculated by Loge(2)/kel. kel was the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Hours | 7.390 (2.5843) | 8.673 (3.3768)

6. Secondary Outcome: Apparent Clearance (CL/F) of PF-07321332 From Plasma
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent clearance) is influenced by the fraction of the dose absorbed. CL/F was calculated as dose/AUCinf.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Liters per hour | 6.812 (31) | 8.148 (36)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07321332
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. Vz/F was calculated as dose/(AUCinf*kel). kel was the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours post-dose on Day 1 of Period 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Liters | 68.77 (41) | 96.88 (38)

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was an AE which resulted in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to maximum of 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 of dosing in the study up to maximum of 35 days after last dose of study drug (approximately maximum of 40 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Participants
  TEAEs | 6 | 5
  SAEs | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Clinical laboratory abnormalities included following criteria: a) hematology evaluation included eosinophils/leukocytes greater than (>) 1.2* upper limit of normal (ULN), monocytes/leukocytes >1.2*ULN; b) clinical chemistry evaluation included urobilinogen greater than or equal to (>=) 1, fibrinogen >1.25*baseline; c) urinalysis evaluation included urine hemoglobin >=1.
Time Frame: Day -1 of Period 1 up to Day 3 of Period 2 (maximum of 8 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Participants | 4 | 4

10. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria for Vital Signs
Description: Vital signs evaluations included supine blood pressure (BP) and pulse rate. The pre specified criteria for vital signs included systolic blood pressure (BP) minimum (min.) less than (<) 90 millimeter of mercury (mmHg); systolic BP change from baseline maximum (max.) decrease >= 30 mmHg, max. increase >=30 mmHg; diastolic BP min. <50mmHg; diastolic BP change from baseline max. decrease >=20, max. increase >=20; supine pulse rate min. <40 beats per minute (bpm) and max. >120 bpm.
Time Frame: Day 1 (pre-dose) of Period 1 up to Day 3 of Period 2 (maximum of 7 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

11. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria for 12-Lead Electrocardiogram (ECG) Values
Description: A 12-lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured PR, QT, and QTc intervals and QRS complex. All scheduled ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position. The pre specified criteria for ECG values included absolute value of QTCF (Fridericia's correction formula): >=450 to less than or equal to (<=) 480 milliseconds, >480 to <=500 milliseconds, >500 milliseconds, increase from baseline >30 - <=60, increase from baseline >60. PR interval: >=300 milliseconds, increase from baseline: baseline >200 milliseconds and max. increase >=25% and baseline <=200 milliseconds and max. increase >=50%; QRS duration: >=140 milliseconds, increase from baseline >=50%.
Time Frame: Day 1 (pre-dose) of Period 1 up to Day 3 of Period 2 (maximum of 7 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dosing in the study up to maximum of 35 days after last dose of study drug (approximately maximum of 40 days)
Arm/Group | PF-07321332 300 mg/Ritonavir 100 mg Fed | PF-07321332 300 mg/Ritonavir 100 mg Fasted
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07321332 300 mg/Ritonavir 100 mg Fed (N=12) | PF-07321332 300 mg/Ritonavir 100 mg Fasted (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Dysgeusia (Nervous system disorders) | 5 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT05129475/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT05129475/SAP_001.pdf